CLINICAL TRIAL: NCT06543914
Title: A ProspeCtive ObseRvatioNal Study of Atogepant Effectiveness in Routine Clinical Practice
Brief Title: Observational Study of Oral Atogepant to Evaluate Real-World Effectiveness in Adult Participants With Migraine
Acronym: CORNERSTONE
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-880
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Migraine
Keywords: Migraine; Atogepant; Qulipta; Aquipta
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Atogepant: Participants will receive atogepant as prescribed by their physician in routine clinical practice.

SUMMARY:
Migraine is a neurological disease characterized by moderate or severe headache, associated with nausea, vomiting, and/or sensitivity to light and sound. This study will evaluate the effectiveness of atogepant in treating adult participants with migraine in a real-world setting.

Atogepant is an approved drug for preventive treatment of migraine in adults. Approximately 1000 adult participants who are prescribed atogepant by their doctors will be enrolled in this study across the world.

Participants will receive atogepant oral tablets as prescribed per standard clinical practice and will be followed for 2 years.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* At least 1-year history of migraine with or without aura consistent with a diagnosis according to the International Classification of Headache Disorders (ICHD)-3, 2018.
* Prescribed atogepant according to the relevant approved local label.
* For participants who initiate atogepant at the prescribing physician or treating health care provider (HCP) discretion as part of their routine clinical care, the decision to administer atogepant must be made prior to and independent of recruitment into the study.
* Willing and able to comply with the requirements of the study.
* Not on concomitant preventive medication for migraine or have been on a stable preventive medication for migraine for at least 3 months prior to enrollment in the study. If on a stable preventive medication, the prescribing physician or treating HCP and participant must confirm that there is no plan to change concomitant preventive medication during the first 12 weeks of the study.

Exclusion Criteria:

* Previously exposed to atogepant as routine therapy or from clinical trials experience prior to entry.
* Contraindications to atogepant as per local labeling.
* Pregnant or planning to be pregnant or women of childbearing potential not using contraception.
* Enrolled in any interventional studies that may include investigational compounds for migraine, or non-AbbVie observational studies.
* In the opinion of the prescribing physician or treating HCP, the participant has a history or current evidence of any condition that might interfere with patient's ability to comply with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with migraine who are prescribed atogepant by their physician per routine standard of care
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a rating of "much better" or "very much better" as assessed by the Patient Global Impression of Change (PGI-C) | Week 12
  PGI-C is a single item used to measure the patient's impression of overall change in migraine since the first dose of atogepant. The measure uses a 7-point rating scale with responses ranging from "very much better" to "very much worse".

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (107):
- United States (12):
  - Neurology and Neurodiagnostics of Alabama /ID# 267614, Hoover, Alabama
  - Rehabilitation & Neurological Services /ID# 267612, Huntsville, Alabama
  - Barrow Neurological Institute - Dignity Health St. Joseph's Hosp and Medical Ctr /ID# 267610, Phoenix, Arizona
  - Kenneth Martinez MD, A Medical Corp /ID# 267834, Aliso Viejo, California
  - Los Angeles Headache Center /ID# 267570, Los Angeles, California
  - Alcanza Clinical Research, LLC /ID# 267838, Lake Mary, Florida
  - Norton Cancer Institute - St. Matthews /ID# 267605, Louisville, Kentucky
  - Dent Neurologic Institute - Amherst /ID# 267606, Amherst, New York
  - Grace Forde /ID# 267596, North New Hyde Park, New York
  - Thomas Jefferson University Hospital /ID# 267572, Philadelphia, Pennsylvania
  - Inova Health Care System /ID# 267615, Falls Church, Virginia
  - Neuroscience Group /ID# 267571, Neenah, Wisconsin
- Belgium (8):
  - Cliniques Universitaires UCL Saint-Luc /ID# 270545, Brussels, Brussels Capital
  - Universitair Ziekenhuis Brussel /ID# 269799, Jette, Brussels Capital
  - Chu Tivoli /ID# 271254, La Louvière, Hainaut
  - Centre Hospitalier Régional de la Citadelle /ID# 270539, Liège, Liege
  - Groupe Sante CHC - Clinique du MontLegia /ID# 270218, Liège, Liege
  - OLV Ziekenhuis Aalst /ID# 270284, Aalst, Oost-Vlaanderen
  - AZ Sint-Jan Brugge /ID# 270540, Bruges, West-Vlaanderen
  - AZ Groeninge /ID# 272772, Kortrijk, West-Vlaanderen
- Canada (10):
  - Calgary Headache Assessment and Management Program /ID# 270266, Calgary, Alberta
  - Burrard Health Center /ID# 270268, Vancouver, British Columbia
  - Dr. Renju Kuriakose Prof. Corp. /ID# 273178, Saint John, New Brunswick
  - Maritime Neurology /ID# 270270, Halifax, Nova Scotia
  - Centricity /ID# 271478, London, Ontario
  - London Health Sciences Centre - Victoria Hospital & Children's Hospital /ID# 270943, London, Ontario
  - Bayshore Neurology /ID# 270673, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre /ID# 273207, Toronto, Ontario
  - Centre de Recherche St-Louis /ID# 270957, Lévis, Quebec
  - Genge Partners /ID# 270267, Montreal, Quebec
- Germany (14):
  - Universitaetsklinikum Heidelberg /ID# 278134, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen /ID# 275762, Tübingen, Baden-Wurttemberg
  - Praxis fur Neurologie Dr. med. Martin Delf /ID# 275918, Hoppegarten, Brandenburg
  - Zentrum Für Klinische Forschung Dr. Irma Schöll /ID# 275642, Bad Homburg, Hesse
  - Evangelisches Krankenhaus Oldenburg /ID# 275823, Oldenburg, Lower Saxony
  - Universitaetsmedizin Greifswald /ID# 276678, Greifswald, Mecklenburg-Vorpommern
  - ZNS Siegen /ID# 275660, Siegen, North Rhine-Westphalia
  - Dres. Huhn-Doll/Siquet/Vocke /ID# 279583, Velbert, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 275759, Dresden, Saxony
  - Schmerzklinik Kiel /ID# 275592, Kiel, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 275760, Berlin
  - Schmerzzentrum Berlin /ID# 275819, Berlin
  - Neurologischen Facharztzentrum Berlin /ID# 275919, Berlin
  - Städtisches Klinikum Brandenburg /ID# 275725, Brandenburg
- Italy (9):
  - IRCCS Ospedale San Raffaele /ID# 273153, Milan, Milano
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli /ID# 275269, Naples, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 274651, Rome, Roma
  - Sapienza University of Rome /ID# 273506, Rome, Roma
  - Azienda Ospedaliero Universitaria delle Marche /ID# 273349, Ancona
  - Policlinico di Bari Ospedale Giovanni XXIII /ID# 275336, Bari
  - Azienda Ospedaliero-Universitaria Renato Dulbecco /ID# 272696, Catanzaro
  - Fondazione Mondino Istituto Neurologico Nazionale a Carattere Scientifico IRCCS /ID# 273155, Pavia
  - Azienda Sanitaria Universitaria Giuliano Isontina - Trieste /ID# 274413, Trieste
- Netherlands (5):
  - Gelre Ziekenhuis /ID# 272429, Apeldoorn, Gelderland
  - Maxima Medisch Centrum, Locatie Veldhoven /ID# 270278, Veldhoven, North Brabant
  - Zaans Medisch Centrum /ID# 269603, Zaandam, North Holland
  - Isala, locatie Zwolle /ID# 269602, Zwolle, Overijssel
  - Maasstad Ziekenhuis /ID# 269601, Rotterdam, South Holland
- Norway (2):
  - Hodeverket /ID# 271383, Sandnes, Rogaland
  - Oslo Hodepinesenter AS /ID# 271384, Oslo
- Portugal (7):
  - Unidade Local de Saude do Alto Ave, EPE /ID# 274767, Guimarães, Braga District
  - Hospital da Luz /ID# 267002, Lisbon, Lisbon District
  - Unidade Local de Saude de Loures-Odivelas, EPE /ID# 274764, Loures, Lisbon District
  - CUF Sintra Hospital /ID# 272394, Sintra, Lisbon District
  - Campus Neurológico Sénior /ID# 272392, Torres Vedras, Lisbon District
  - Hospital CUF Coimbra /ID# 272393, Coimbra
  - Hospital CUF Porto /ID# 272788, Porto
- Spain (13):
  - Hospital Regional Universitario de Malaga /ID# 268272, Málaga, Andalusia
  - Hospital Universitari de Bellvitge /ID# 268224, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Severo Ochoa /ID# 268249, Leganés, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 268246, Majadahonda, Madrid
  - Hospital Universitario Central de Asturias /ID# 276477, Oviedo, Principality of Asturias
  - Hospital Universitario Virgen Macarena /ID# 268244, Seville, Sevilla
  - Hospital Universitario Vall de Hebron /ID# 268222, Barcelona
  - Hospital Universitario de La Princesa /ID# 268245, Madrid
  - Hospital Universitario La Paz /ID# 268238, Madrid
  - Hospital Alvaro Cunqueiro /ID# 268248, Pontevedra
  - Hospital Universitario Virgen del Rocio /ID# 268223, Seville
  - Hospital Clinico Universitario de Valladolid /ID# 268225, Valladolid
  - Hospital Clinico Universitario Lozano Blesa /ID# 268243, Zaragoza
- Sweden (3):
  - Karolinska Universitetssjukhuset - Huddinge /ID# 265295, Huddinge, Stockholm County
  - Neurology Clinic /ID# 266707, Stockholm, Stockholm County
  - Skaneuro /ID# 265203, Lund
- Switzerland (10):
  - NeuroPraxis Birseck /ID# 266140, Reinach, Basel-Landschaft
  - ZURZACH Care /ID# 265697, Bad Zurzach, Canton of Aargau
  - CHUV, Centre hospitalier universitaire vaudois /ID# 266551, Lausanne, Canton of Vaud
  - Kopfwehzentrum Hirslanden Zuerich /ID# 265817, Zollikon, Canton of Zurich
  - Neurozentrum Bellevue /ID# 277666, Zurich, Canton of Zurich
  - University Hospital Zurich /ID# 276450, Zurich, Canton of Zurich
  - DYA Swiss Institut SA /ID# 266891, Lugano, Canton Ticino
  - EOC Ospedale Regionale Lugano /ID# 266887, Lugano, Canton Ticino
  - Hôpital De Sion /ID# 276360, Sion, Valais
  - Inselspital, Universitaetsspital Bern /ID# 265818, Bern
- Taiwan (2):
  - Tri-Service General Hospital /ID# 272082, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 272084, Taoyuan
- American Center of Neurology and Psychiatry /ID# 276429, Abu Dhabi, United Arab Emirates
- United Kingdom (11):
  - Hull Royal Infirmary /ID# 276819, Hull, East Riding Of Yorkshire
  - Western General Hospital - NHS Lothian /ID# 277029, Edinburgh, Edinburgh, City of
  - Guy's Hospital /ID# 276817, London, Greater London
  - King'S College Hospital /ID# 276818, London, Greater London
  - Cripps Health Centre /ID# 277474, Nottingham, Nottinghamshire
  - University Hospitals North Midlands - Royal Stoke University Hospital /ID# 276821, Stoke-on-Trent, Staffordshire
  - Leeds Teaching Hospitals NHS Trust /ID# 279417, Leeds, West Yorkshire
  - Great Western Hospital /ID# 276693, Swindon, Wiltshire
  - Worcestershire Royal Hospital /ID# 276902, Worcester, Worcestershire
  - Ulster Hospital - South Eastern Health & Social Care Trust /ID# 276900, Belfast
  - University Hospital of Wales /ID# 276822, Cardiff

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-880